CLINICAL TRIAL: NCT03271073
Title: A Exploratory Study of Apatinib in Combination With S1 in Patients With Advanced Gastric Evaluating the Efficacy and Safety
Brief Title: A Study of Apatinib Combined With S1 in Patients With Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, assistant dean, professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-Y001
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; gastroesophageal junction cancer; Apatinib; S1
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; S 1 (combination)

ARMS (1):
- Apatinib plus S1 (Experimental): patients with advanced gastric cancer enrolled after failure of first-line systemic chemotherapy will be given Apatinib plus S1 till progressive disease,death or non-tolerable toxicity
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib,500mg,qd,po,d1-21;S1,40mg,bid,d1-14;every 21days a cycle
  Other Names: S1

SUMMARY:
Antiangiogenesis therapy plays an important role in cancer treatment. Apatinib showed good safety and efficacy as third-line therapy for advanced gastric cancer.We conducted this trial to investigate the safety and efficacy of apatinib combined with S1 after failure of first-line chemotherapy in advanced gastric cancer or gastroesophageal junction carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, aged between 18 and 75 years old;
2. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2;
3. Histologically confirmed advanced or metastatic adenocarcinoma of gastric cancer(AGC) , including adenocarcinoma of the gastroesophageal junction ,one or more measurable or nonmeasurable evaluable lesions per RECIST 1.1;
4. Failure or intolerance to at least one prior line of systemic chemotherapy regimen;
5. Adequate liver, renal, heart, and bone-marrow functions ( hemoglobin≥ 80g/L, platelets ≥ 100 × 10*9/L, neutrophil ≥1.5 × 10*9/L, total bilirubin ≤1.5 ×ULN, and serum transaminase≤2.5×ULN);
6. Expected survival of ≥ 12 weeks.

Exclusion Criteria:

1. Subjects with poor-controlled arterial hypertension (systolic blood pressure> 140 mmHg and diastolic blood pressure > 90 mm Hg) despite standard medical management; Coronary heart disease greater than ClassI; I-level arrhythmia (including QT interval prolongation, for man ≥ 450 ms, for woman ≥ 470 ms) together with Class I cardiac dysfunction;
2. Subjects with high gastrointestinal bleeding risk, including the following conditions: local active ulcer lesions with positive fecal occult blood test (++); history of black stool, or vomiting blood in the past 2 months;
3. Abnormal Coagulation (INR>1.5、APTT>1.5 UNL), with tendency of bleed;
4. Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
5. Previous treatment with VEGFR inhibitor (i.e. Apatinib, sorafenib, sunitinib);
6. With psychotropic drug abuse history and can't get rid of or mental disorder patients;
7. Associated with CNS (central nervous system) metastases;
8. Active bacterial infections;
9. Pregnant or breast-feeding women;
10. Any other condition that might place the patient at undue risk or preclude a patient from completing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 1 year
  defined as the time from randomize to progression or death; RECIST guidelines were used to define all responses after patients had received every 6 weeks of therapy

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately 2 years
  defined as the time from randomize to death
Safety (incidence of adverse events) | Approximately 1 year
  incidence of adverse events
Quality of life(QoL) | Approximately 2 years
  as measured by the European Organization for Research and Treatment of Cancer questionnaire (EORTC QLQ C30)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Deng, M.D., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No